CLINICAL TRIAL: NCT00634426
Title: Surgical Versus Nonoperative Treatment of Metastatic Epidural Spinal Cord Compression. Quality of Life and Cost-effectiveness Outcomes
Brief Title: Surgical Versus Nonoperative Treatment of Metastatic Epidural Spinal Cord Compression
Acronym: MESCC
Status: Completed | Type: Observational
Sponsor: AOSpine North America Research Network (Network)
Collaborators: AOSpine North America (Industry)
Responsible Party: Sponsor
Other Study IDs: 1011
Record Dates: First submitted 2008-03-03; First posted 2008-03-13 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Epidural Spinal Cord Compression
Keywords: Spine; Neoplasm metastasis; Treatment, surgical; Treatment, nonoperative; Quality of life
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: De novo surgical cohort
  Interventions: Procedure: Surgical excision of the metastatic process
- 2: Nonoperative treatment cohort
  Interventions: Radiation: Radiotherapy of the metastatic spine process
- 3: Secondary surgical treatment cohort
  Interventions: Procedure: Surgical excision of the metastatic process

INTERVENTIONS:
Procedure: Surgical excision of the metastatic process — Surgical excision of the metastatic process
  Groups: 1; 3
Radiation: Radiotherapy of the metastatic spine process — Standard of care radiotherapy for patients with metastatic epidural spinal cord compression.
  Groups: 2

SUMMARY:
The aim of this trial is to evaluate the differences in pain relief, neurological function, quality of life and survival in patients with metastatic epidural spinal cord compression (MESCC) who are managed with a combination of surgery and radiotherapy versus radiotherapy alone.

Further we shall evaluate cost-effectiveness of the two treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Single symptomatic metastatic epidural spinal compression at any level confirmed by MRI
* Age 18 and more
* Able and willing to give written informed consent to participate in the study
* Able to read and write English on an elementary level

Exclusion Criteria:

* Multiple symptomatic spinal metastases
* Radiosensitive tumors
* Radioresistant tumors
* Primary cancer site in CNS or spine
* Poor life expectancy (< 3 months)
* Patients with a tumor that has compressed only the cauda equina or spinal roots
* Has a recent history of substance abuse
* Is a prisoner
* Currently involved in another study
* has a disease or condition that would preclude accurate evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present for the treatment of new (cohorts 1 & 3) or old (cohort 2) metastatic epidural spinal cord compression at the participating sites.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2008-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in spine-associated pain intensity (BPI) measured by Brief Pain Inventory | 6 weeks / 3, 6, 9, 12, 18, 24 months
Neurological outcomes measured by American Spinal Injury Association (ASIA) Motor Scale structured clinical examination | 24 months

SECONDARY OUTCOMES:
Survival | 24 months
SF-36 v2 | 24 month
EQ-5D | 24 months
Oswestry Disability Index (ODI) | 24 months
Caregiver Activity Survey | 24 months
Adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fehlings, MD FRCSC, Principal Investigator — University of Toronto
Locations (10):
- United States (7):
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University and The Rothman Institute, Philadelphia, Pennsylvania
  - University of Texas Hospital / MD Anderson Cancer Center, Houston, Texas
  - West Viginia University, Morgantown, West Virginia
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - University of Toronto, Toronto, Ontario

REFERENCES:
- [Background] Sciubba DM, Petteys RJ, Dekutoski MB, Fisher CG, Fehlings MG, Ondra SL, Rhines LD, Gokaslan ZL. Diagnosis and management of metastatic spine disease. A review. J Neurosurg Spine. 2010 Jul;13(1):94-108. doi: 10.3171/2010.3.SPINE09202. PMID 20594024
- [Background] Furlan JC, Chan KK, Sandoval GA, Lam KC, Klinger CA, Patchell RA, Laporte A, Fehlings MG. The combined use of surgery and radiotherapy to treat patients with epidural cord compression due to metastatic disease: a cost-utility analysis. Neuro Oncol. 2012 May;14(5):631-40. doi: 10.1093/neuonc/nos062. Epub 2012 Apr 14. PMID 22505658
- [Result] Fitzpatrick D, Grabarz D, Wang L, Bezjak A, Fehlings MG, Fosker C, Rampersaud R, Wong RK. How effective is a virtual consultation process in facilitating multidisciplinary decision-making for malignant epidural spinal cord compression? Int J Radiat Oncol Biol Phys. 2012 Oct 1;84(2):e167-72. doi: 10.1016/j.ijrobp.2012.03.057. Epub 2012 Jun 8. PMID 22682804
- [Result] Fisher CG, Schouten R, Versteeg AL, Boriani S, Varga PP, Rhines LD, Kawahara N, Fourney D, Weir L, Reynolds JJ, Sahgal A, Fehlings MG, Gokaslan ZL. Reliability of the Spinal Instability Neoplastic Score (SINS) among radiation oncologists: an assessment of instability secondary to spinal metastases. Radiat Oncol. 2014 Mar 4;9:69. doi: 10.1186/1748-717X-9-69. PMID 24594004
- [Result] Fisher CG, Versteeg AL, Schouten R, Boriani S, Varga PP, Rhines LD, Heran MK, Kawahara N, Fourney D, Reynolds JJ, Fehlings MG, Gokaslan ZL. Reliability of the spinal instability neoplastic scale among radiologists: an assessment of instability secondary to spinal metastases. AJR Am J Roentgenol. 2014 Oct;203(4):869-74. doi: 10.2214/AJR.13.12269. PMID 25247954